CLINICAL TRIAL: NCT02099084
Title: Acute Effects of a Glucagon-like Peptide 2 Analog, Teduglutide, on Gastrointestinal Motor Function and Permeability in Patients With Short Bowel Syndrome on Home Parenteral Nutrition
Brief Title: Short Bowel Syndrome and Teduglutide Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, Primary Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-004866; UL1TR000135 (NIH)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teduglutide First, then Placebo (Experimental): Teduglutide 0.05 mg/kg/d administered subcutaneously for 7 days, followed by a 14-day washout period, and placebo administered subcutaneously for 7 days.
  Interventions: Drug: Teduglutide; Drug: Placebo
- Placebo First, then Teduglutide (Placebo Comparator): Placebo administered subcutaneously for 7 days, followed by a 14-day washout period, and Teduglutide 0.05 mg/kg/d administered subcutaneously for 7 days.
  Interventions: Drug: Teduglutide; Drug: Placebo

INTERVENTIONS:
Drug: Teduglutide — Participants will receive Teduglutide 0.05 mg/kg/d administered subcutaneously.
  Other Names: Gattex; Revestive
Drug: Placebo — Participants will receive placebo matching study drug, administered subcutaneously.

SUMMARY:
This research study was done to see what the effects are of Teduglutide on people with short bowel syndrome (SBS). Teduglutide is a synthetic medication administered as an injection, which has shown to increase intestinal blood flow, inhibit gastric secretion, increase growth of intestinal cells and increase absorption of nutrients. Teduglutide has demonstrated to decrease Total Parenteral Nutrition (TPN) requirements by 20%. Teduglutide is approved by the Food and Drug Administration (FDA) for the treatment of adult patients with Short Bowel Syndrome (SBS) who are dependent on parenteral support.

The primary hypotheses for this study were 1) that Teduglutide significantly increases the gastric emptying half time of solids when compared to placebo. 2) Teduglutide will significantly decrease the intestinal permeability and urinary excretion of lactulose when compared to placebo.

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) refers to the anatomical and/or functional decrease in small intestinal absorptive capacity, mostly caused by extensive intestinal resections. The decrease in intestinal absorptive capacity leads to malabsorption causing malnutrition, dehydration and weight loss, all of which severely impact patient's quality of life.

In this study, qualifying participants were assigned to 2 different treatment arms consisting of placebo or Teduglutide 0.05 mg/kg subcutaneously daily for seven days. Subsequently, participants were switched over to the alternate treatment arm for seven days, after a washout period of at least seven days. In both arms, after six days of treatment or placebo, participants underwent a series of measurements during day 7 of treatment, including 8 hour GI transit, permeability measurements by using mannitol and lactulose (0-2h, 2-8h collections), and 8 hour urine and stool collections for measurement of volume. Throughout the study participants filled out a food diary and a stool diary (number, consistency, ease of passage) every day.

On day 7 of each intervention period participants arrived in the clinical research unit after having fasted for at least 8 hours. Women of childbearing potential had a pregnancy test. Participants then received their seventh dose of placebo or Teduglutide (1 dose, 1 hour before breakfast). Technetium sestamibi (99mTc) pellets were ingested in a scrambled egg, toast, and milk meal (218 kcal) to facilitate measurement of gastric transit. All subjects received a standard 550 kcal meal at 4 hours (chicken meal) after the radiolabeled meal.

ELIGIBILITY:
Inclusion criteria:

* Short bowel syndrome
* Dependent on parenteral nutrition

Exclusion criteria:

* Pregnant, trying to become pregnant or lactating
* Diabetes
* Alcohol or drug abuse within the last year by history
* Active Crohn's disease as evaluated by standard procedures employed by the investigator
* History of radiation enteritis, scleroderma, celiac disease, tropical sprue, diabetes, chronic pseudo-obstruction or malignancies
* Previous use of Teduglutide or potential allergies to Teduglutide or its constituents
* Any hospitalization within 1 month before screening
* Use of Octreotide, intravenous glutamine growth hormone or growth factors such as native Glucagon-like Peptide 2 (GLP-2) within the last 12 weeks
* Infliximab or other biological agents, Azathioprine, Methotrexate, Cyclosporine, Tacrolimus, Sirolimus, should be stable for at least 8 weeks prior to baseline and remain stable during the study

  - Any investigational drug within last 30 days
* Diuretics and oral rehydration solutions will be required to be stable for ≥4 weeks prior to baseline evaluations and remain stable during the study
* Change in dose of antimotility or secretory agents from 2 days prior to, and throughout the two phases and washout periods of the study
* Use of tobacco products within the prior 1 month (since nicotine can affect permeability)
* Use of NSAIDS or aspirin within the past week
* Use of oral corticosteroids within the previous 6 weeks
* Ingestion of artificial sweeteners such as Splenda (sucralose), Nutrasweet (aspartame), lactulose or mannitol 2 days each of the study measurement days, e.g., foods to be avoided are sugarless gums or mints and diet soda
* History of pancreatitis
* Primary renal impairment (estimated glomerular filtration rate (eGFR)) <30 ml/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iturrino J, Camilleri M, Acosta A, O'Neill J, Burton D, Edakkanambeth Varayil J, Carlson PJ, Zinsmeister AR, Hurt R. Acute Effects of a Glucagon-Like Peptide 2 Analogue, Teduglutide, on Gastrointestinal Motor Function and Permeability in Adult Patients With Short Bowel Syndrome on Home Parenteral Nutrition. JPEN J Parenter Enteral Nutr. 2016 Nov;40(8):1089-1095. doi: 10.1177/0148607115597644. Epub 2015 Jul 28. PMID 26223941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic Home Parenteral Nutrition program in Rochester, Minnesota.
Period: First Intervention
Arm/Group | Teduglutide First, Then Placebo | Placebo First, Then Teduglutide
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Washout Period of 14 Days
Arm/Group | Teduglutide First, Then Placebo | Placebo First, Then Teduglutide
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Teduglutide First, Then Placebo | Placebo First, Then Teduglutide
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive placebo first and Teduglutide first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying Half-Time (T1/2)
Description: The time for half of the ingested solids or liquids to leave the stomach.
Time Frame: approximately 2 hours after radiolabeled meal is ingested
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Teduglutide: Teduglutide 0.05 mg/kg/d administered subcutaneously for 7 days in either first intervention period or second intervention period
- Placebo: Placebo administered subcutaneously daily for 7 days in either first intervention period or second intervention period
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
minutes | 113 (16) | 106 (20)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Level of significance = .05; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

2. Secondary Outcome: Change in Small Intestinal and Colonic Permeability as Measured by Urinary Excretion of Mannitol
Description: Permeability is measured through differential excretion of urine saccharides. A sugar solution (200 mg of mannitol and 1 g lactulose in 30 mL of water) was administered with the radiolabeled test meal at visits 1 and 2. Urine was collected during 0-2 and 2-8 hours. A baseline urine sample was also collected prior to ingestion of the sugars. Chemical analysis was preformed with high-speed liquid chromatography tandem mass spectrometry.
Time Frame: baseline, approximately 2 hours and 8 hours after ingestion of radiolabeled meal
Measure: Mean (Standard Error); unit: mg
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
mg
  0 - 2 hours | 16.2 (3.6) | 11.3 (2.2)
  0 - 8 hours | 48.8 (8.9) | 32.7 (5.9)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Comparison between the groups for change between 0- and 2-hours. Level of significance = .05; Test type: Superiority or Other; p = 0.20, t-test, 2 sided
Statistical Analysis 2: Comparison: Teduglutide vs Placebo; Comparison between the groups for change between 0- and 8-hours. Level of significance = .05; Test type: Superiority or Other; p = 0.17, t-test, 2 sided

3. Primary Outcome: Overall Gut Transit
Description: Given the variable extent of the residual length of the small intestine and colon, the proportion emptied from the body at 6 hours was assessed as an overall estimate of the whole gut transit. The 6-hour values for intra-abdominal counts were then compared with the 100% reference values of counts (at time zero, which is immediately after ingestion of the radiolabeled meal) to determine the percentage of isotope retained in the abdomen. 100% minus the percentage of retained isotope reflected the amount emptied from the GI tract.
Time Frame: baseline, approximately 6 hours after ingestion of radiolabeled meal
Measure: Mean (Standard Deviation); unit: Percentage of isotope emptied
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
Percentage of isotope emptied | 53.4 (15) | 62.4 (15.2)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Level of significance = .05; Test type: Superiority or Other; p = 0.075, t-test, 2 sided

4. Secondary Outcome: Change in Small Intestinal and Colonic Permeability as Measured by Urinary Excretion of Lactulose at 2 Hours
Description: as for outcome 2
Time Frame: baseline, approximately 2 hours after ingestion of radiolabeled meal
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
mg | 0.42 (0.14) | 0.38 (0.14)

5. Secondary Outcome: Change in Small Intestinal and Colonic Permeability as Measured by Lactulose/Mannitol Ratio at 2 Hours
Description: as for outcome 2
Time Frame: baseline, approximately 2 hours after ingestion of radiolabeled meal
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
ratio | 0.024 (0.005) | 0.021 (0.005)

6. Other Pre Specified Outcome: Stool Weight at 8 Hours
Description: After an overnight fast, subjects received a single dose of placebo or Teduglutide 1 hour before breakfast, then consumed a radiolabeled meal. After 8 hours a stool collection was taken.
Time Frame: approximately 8 hours after ingestion of radiolabeled meal
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
g | 77 (18) | 106 (43)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Level of significance = .05; Test type: Superiority or Other; p = 0.42, t-test, 2 sided

7. Other Pre Specified Outcome: Urine Volume at 8 Hours
Description: After an overnight fast, subjects received a single dose of placebo or Teduglutide 1 hour before breakfast, then consumed a radiolabeled meal. Urine was collected twice: from the start of the ingestion of the meal to 2 hours, and 2-8 hours. The total volume of urine collected was the sum of these two collections.
Time Frame: Start of the ingestion of the radiolabeled meal until 8 hours after the meal
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 8
mL | 408.9 (52.2) | 365.7 (57.3)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Level of significance = .05; Test type: Superiority or Other; p = 0.34, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 21 days.
Description: Adverse events were recorded in the daily stool diary. Participants were contacted on day 2 and day 5 of each phase of the study medications. Participants also met with study staff on visits 1-3.
Arm/Group | Teduglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=8) | Placebo (N=8)
Moderate abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Headache (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increase in size of stoma (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes